CLINICAL TRIAL: NCT04267796
Title: Reducing Breast Cancer Risk Through Modifying Body Composition and Decreasing Inflammation in Normal Weight Women
Brief Title: Lifestyle Intervention for the Reduction of Breast Cancer Risk in Normal Weight Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Foundation for Women's Cancers (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-0634; NCI-2019-07636 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0634 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-26; First posted 2020-02-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise; Diet Therapy; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (lifestyle intervention) (Experimental): Participants complete lifestyle intervention consisting of 1-3 sets of high-resistance circuit training sessions per week, up to 150 minutes of aerobic training per week, and diet recommendations from a health coach or registered dietitian twice per week for 16 weeks.
  Interventions: Other: Aerobic Exercise; Other: Dietary Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Resistance Training
- Group II (wait-list, lifestyle intervention) (Active Comparator): Participants are placed on a wait-list and then complete lifestyle intervention after 4 months.
  Interventions: Other: Aerobic Exercise; Other: Dietary Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Resistance Training

INTERVENTIONS:
Other: Aerobic Exercise — Complete aerobic training
  Other Names: Aerobic Activity
Other: Dietary Intervention — Receive diet recommendations from health coach or registered dietitian
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Resistance Training — Complete high-resistance circuit training sessions
  Other Names: Strength Training

SUMMARY:
This trial studies how well a lifestyle intervention works in reducing breast cancer risk through changing body composition and decreasing inflammation in normal weight women. This trial may help researchers learn more about diet and exercise programs designed to decrease body fat in postmenopausal women who are of normal weight but have an elevated risk of breast cancer because of excess body fat.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the feasibility of a diet and exercise intervention to decrease body fat in postmenopausal women with normal body mass index (BMI) but high body fat (trunk fat mass 9.4 kg, the 50th percentile of normal BMI women in the Women's Health Initiative [WHI]).

SECONDARY OBJECTIVE:

I. Assess preliminary efficacy of the intervention by evaluating the post-intervention differences between the intervention and control groups in:

IIa. Circulating markers of inflammation and metabolic dysfunction linked to both excess adiposity and breast cancer (high sensitivity C-reactive protein [hsCRP], fasting insulin, leptin, IL-6, triglycerides, sex hormone binding globulin [SHBG], adiponectin, and high density lipoprotein [HDL] cholesterol).

IIb. Body composition body fat, trunk fat mass, fat mass, lean mass, fat-free mass).

EXPLORATORY OBJECTIVE:

I. Exploratory outcomes include fitness (oxygen consumption VO2 peak, sit-to-stand test), behavior (physical activity, energy intake, macronutrient consumption), and quality of life (global health-related quality of life, physical functioning, sleep, menopausal symptoms).

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I: Participants complete lifestyle intervention consisting of 1-3 sets of high-resistance circuit training sessions per week, up to 150 minutes of aerobic training per week, and diet recommendations from a health coach or registered dietitian twice per week for 16 weeks.

GROUP II: Participants are placed on a wait-list and then complete lifestyle intervention after 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-69 years old
* Postmenopausal woman (absence of menstruation for at least one year, or history of bilateral oophorectomy)
* Self-reported height and weight indicating a BMI >= 18.5 and < 25 kg/m^2
* No contraindications to exercise (either no positive responses on the Physical Activity Readiness Questionnaire, or clearance from a health care provider certifying that the participant is healthy enough to exercise)
* No history of invasive cancer, other than non-melanoma skin cancer
* No history of renal disease
* Able to walk without an assistive device
* Not within 3 months of major surgery
* Able to speak/read/write in English
* Has internet access on a computer or mobile device
* A trunk fat mass >= 9.4 kg as indicated by a dual x-ray absorptiometry (DXA) scan
* Height and weight indicating a BMI of >= 18.5 and < 25 kg/m^2 verified at the screening visit

Exclusion Criteria:

* MD Anderson employees that report to the principal investigator of this study
* Participants that cannot engage in the exercise program for more than three weeks during the study period
* Participants that are currently doing strength exercises that work all major muscle groups (defined as: participants who complete more than 16 repetitions per exercise in their current resistance training regimen, or who don't find their last 1-2 reps to be difficult in their current regimen, or who increase the weight in their current routine).

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of a diet intervention to decrease body fat in postmenopausal women with normal BMI but high body. fat. | up to 16 weeks
  Will assessed by the calculated rates, frequencies, and 95% confidence intervals (CIs) for these measures
Evaluate the exercise intervention to decrease body fat in postmenopausal women with normal BMI but high body. fat. | up to 16 weeks
  Will assessed by the calculated rates, frequencies, and 95% confidence intervals (CIs) for these measures

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Basen-Engquist, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org